CLINICAL TRIAL: NCT01859338
Title: Clinical Evaluation of Soft Tissue Detection on MRI, Cone Beam CT and Fan Beam CT and Integration of Functional MR Imaging Into Radiotherapy Planning
Brief Title: Soft Tissue Detection on MRI, Cone Beam CT and Fan Beam CT and Integration of Functional MRI
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM13777; NCI-2013-00847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-13777 (Other: Massey Cancer Center)
Record Dates: First submitted 2013-05-07; First posted 2013-05-21 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer; Prostate Cancer
MeSH Terms: conditions — Lung Neoplasms; Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI, CBCT, FBCT: Patients undergo MRI and fan beam CT (FBCT) at baseline, within the first 3 weeks of radiotherapy and between week 4 and 6 of radiotherapy. Patients with lung cancer may undergo 4D cone beam x-ray CT (CBCT) on the same day as the second and third MRI and FBCT.
  Interventions: Radiation: cone-beam computed tomography; Radiation: magnetic resonance imaging; Radiation: computed tomography

INTERVENTIONS:
Radiation: cone-beam computed tomography — Undergo CBCT
  Other Names: CBCT
Radiation: magnetic resonance imaging — Undergo MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Radiation: computed tomography — Undergo fan beam computed tomography
  Other Names: tomography, computed

SUMMARY:
This clinical trial studies magnetic resonance imaging (MRI), cone beam computed tomography (CT), and fan beam CT in detecting soft tissue in patients with prostate and lung cancer undergoing radiation therapy. Comparing results of diagnostic procedures done before and during radiation therapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the technical feasibility of MRI for performing functional soft-tissue targeting of radiotherapy in the pelvis and thorax. (Group I) II. Acquire clinical MR imaging data to evaluate image quality tradeoffs and operational parameter settings. (Group I) III. Validate the selection of MRI technique factors by comparing visibility of soft tissue structures in MRIs, cone beam (CB)CTs and fan beam (FB)CTs of the same patient. (Group II) IV. Assess the feasibility of using deformable image registration to map contours from FBCT to MRI, CBCT to MRI, MRI to MRI and vice versa. (Group II) V. Compare morphologic and functional changes in target and normal structures, visualized on MRI, CBCT and FBCT images, in response to radiation therapy and identify opportunities for treatment adaptation. (Group II)

OUTLINE:

Patients undergo MRI and FBCT at baseline, within the first 3 weeks of radiotherapy and between week 4 and 6 of radiotherapy. Patients with lung cancer may undergo 4 dimensional (4D) CBCT on the same day as the second and third MRI and FBCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung cancer visible on CT who are scheduled to receive radiation treatment to the area of the primary tumor will be eligible for this study - Renal function tests (blood urea nitrogen [BUN], creatinine [Cr], glomerular filtration rate [GFR]) within 30 days of MRI with GFR > 59 mL/min
* All patients must give written informed consent on a form that includes Health Insurance Portability and Accountability Act (HIPAA) authorization; patient therapy will not be directed by enrollment in this study; participation in this study will not preclude patient participation in additional therapy protocols; subjects will all be recruited from patients undergoing radiotherapy at one of the Virginia Commonwealth University (VCU)-affiliated radiotherapy clinics

Exclusion Criteria:

* Patients requiring continuous supplemental oxygen
* Patients with metal implants including pace makers and defibrillators
* Patients with cerebral aneurysm clips or middle ear implant
* Patients with pain pump, a programmable shunt, or non-surgical metal (i.e. a foreign body)
* Claustrophobic patients
* Prior radiotherapy to body area under investigation
* No vulnerable populations will be enrolled (prisoners, children, pregnant females, or institutionalized individuals); women of childbearing potential will undergo a pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated in the Massey Cancer Center Radiation Therapy will be recruited for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-03-06; Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Technical feasibility of MRI for performing functional soft-tissue targeting of radiotherapy in the pelvis and thorax | up to 6 weeks
  Make a preliminary comparison of soft tissue structures delineated from MRI to those identified based on cone beam CT (CBCT) and fan beam CT (FBCT). In addition, variations in the soft tissue identification from repeated MR imaging will be compared to morphological imaging.
Clinical MR imaging data in evaluating image quality tradeoffs and operational parameter settings | Up to 6 weeks
  Image quality will be assessed by evaluating the utility of various comparative image quality quantifiers such as signal-to-noise ratio (SNR), resolution, and reproducibility of soft-tissue structure identification.

SECONDARY OUTCOMES:
Visibility of soft tissue structures in MRIs, CBCTs and FBCTs of the same patient | Up to 6 weeks
  Compared using a paired t-test.
Deformable image registration to map contours from FBCT to MRI, CBCT to MRI, MRI to MRI and vice versa | Up to 6 weeks
  Compared using a paired t-test.
Functional changes in target and normal structures, visualized on MRI, CBCT and FBCT images, in response to radiation therapy and identify opportunities for treatment adaptation | Up to 6 weeks
  Compared using a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Weiss, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States